CLINICAL TRIAL: NCT00281502
Title: The Role of Bacterial Overgrowth and Delayed Intestinal Transit in Hepatic Encephalopathy. Phase A: Breath Testing and Colonic Transit in Hepatic Encephalopathy. Phase B: A Randomized Double Blind, Placebo Controlled Trial of Rifaximin for Hepatic Encephalopathy
Brief Title: The Role of Bacterial Overgrowth and Delayed Intestinal Transit in Hepatic Encephalopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sam Sigal, Weill Medical College of Cornell University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Salix-RifaxPSE-BactOvrGrwth-01
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Hepatic Encephalopathy; Hepatitis C; Liver Cirrhosis
Keywords: Hepatic Encephalopathy; Hepatitis C; Liver Cirrhosis; Bacterial Overgrowth
MeSH Terms: conditions — Hepatic Encephalopathy; Hepatitis C; Liver Cirrhosis | interventions — Rifaximin; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rifaximin (drug) — Rifaximin 400mg three (3) times daily
  Other Names: Xifaxan

SUMMARY:
The study will be conducted in two phases. Phase A will evaluate the contribution of bacterial overgrowth and colonic inertia to development of Hepatic Encephalopathy (HE)in 50 ambulatory subjects with HE and hepatitis C cirrhosis. This phase will include a Screening and Evaluation Visit.

Phase B will evaluate the effect of rifaximin on bacterial outgrowth and severity of HE in 20 of the subjects enrolled in Phase A who have a somewhat greater degree of encephalopathy.

The purpose of this study is to evaluate the following:

1. the relationship between bacterial overgrowth and the presence and severity of HE in patients with hepatitis C cirrhosis;
2. the effectiveness and tolerability of rifaximin relative to placebo in treatment of HE associated with hepatitis C cirrhosis;
3. the relationship between bacterial overgrowth and the presence and severity of HE before and after rifaximin treatment.

DETAILED DESCRIPTION:
Hepatic encephalopathy is a frequent and occasionally refractory complication of cirrhosis and is associated with impaired quality of life. Its severity may not correlate with other parameters of liver dysfunction. Although multiple pathogenic mechanisms for the condition have been proposed, most include the participation of bacterial toxins, especially ammonia, produced in the gastrointestinal tract. Treatment options for hepatic encephalopathy at this time are limited to lactulose and neomycin. Lactulose is frequently poorly tolerated, and many patients are non-compliant with its use. In patients with renal insufficiency in whom hepatic encephalopathy is frequently problematic, use of neomycin is contraindicated due to ototoxicity and nephrotoxicity.

Autonomic dysfunction is common in patients with cirrhosis and could contribute to the development of hepatic encephalopathy by impairment of intestinal motility, leading to bacterial overgrowth and colonic inertia.

The following questions will be addressed:

A. Is impaired intestinal transit and bacterial overgrowth associated with the presence and severity of hepatic encephalopathy?

50 patients will undergo a detailed clinical evaluation for severity of liver disease, hepatic encephalopathy and assessment of intestinal transit and bacterial overgrowth with radiographic marker study and breath test analysis. Multivariate analysis will then be performed to determine the relationship of intestinal transit and evidence of bacterial overgrowth with the presence and severity of hepatic encephalopathy.

B. Does treatment with rifaximin improve bacterial overgrowth and hepatic encephalopathy?

20 patients from the above population with significant encephalopathy will be randomized to receive either rifaximin or placebo. Post-treatment evaluation for severity of hepatic encephalopathy and breath test analysis for bacterial overgrowth will then be performed. The effect of treatment on changes in hepatic encephalopathy and bacterial overgrowth and the relationship between changes in bacterial overgrowth and severity of hepatic encephalopathy will also be assessed.

Phase A Endpoints: Degree of bacterial overgrowth and its correlation with the grade of hepatic encephalopathy (if present).

Phase B Endpoints: To demonstrate improvement in degree of HE with treatment of Rifaximin

Efficacy Endpoints The primary efficacy endpoint for Phase B of the study will be the change from baseline in the proportion of patients with no HE, minimal HE (no symptoms, abnormal psychometric testing), mild persistent HE (mild symptoms), and persistent Stage II HE (presence of asterixis, history of hospitalization for spontaneous Stage III or IV HE).

Secondary efficacy endpoints for Phase B will be the following:

To demonstrate improvement in intestinal transit time for patients (based on Lactulose Hydrogen Breath Test) To demonstrate improvement in bacterial overgrowth, improved insomnia, flatulence, and quality of life.

To demonstrate that rifaximin improved patients' symptoms of insomnia, flatulence, and quality of life measure with the degree of bacterial overload and the impaired intestinal transit time.

ELIGIBILITY:
Phase A Inclusion Criteria:

* Subject is 18 to 70 years of age, inclusive.
* Subject has cirrhosis due to chronic HCV infection as documented by:
* Subject has evidence of hepatic encephalopathy as evidenced by:
* Neuro-psychometric Testing (Number Connection Test, Trails Test, etc.)
* Subject is non-azotemic (creatinine <1.5mg/dL) and ambulatory at screening.
* Subject has cirrhosis due to chronic HCV as documented by: pathologic or clinical and radiographic evidence of cirrhosis with a positive HCV RNA PCR level.

Phase A Exclusion Criteria:

* Subject has received active interferon therapy within 2 weeks of enrollment.
* Subject is pregnant or lactating.
* Subject has a life expectancy of less than 100 days.
* Subject has a history of alcohol abuse within 6 months of enrollment.
* Subject has active gastrointestinal bleeding at time of enrollment.
* Subject has used an agent that alters intestinal motility, eg, methadone, cholestyramine, tricyclic antidepressants.
* Subject is unable to take oral medication.
* Subject has used neomycin or other antibiotic within 2 weeks of enrollment or is actively using lactulose at time of enrollment.
* Subject is taking or has hypersensitivity or allergy to rifaximin or rifampin.
* Subject requires long term antibiotic therapy (eg, Lyme Disease, tuberculosis).
* Subject has known or suspected alcohol abuse or illicit drug use within 1 year of enrollment.
* Subject has participated in an investigational drug or device study within the 30 days prior to randomization.
* Subject has received rifaximin within the last 30 days.
* Subject has concomitant disease or condition that could interfere with, or for which treatment could interfere with the conduct of the study, or could in the opinion of the investigator increase the risk of AEs for the subject's participation in the study.
* Subject is unwilling or unable to comply with the study protocol for any other reason.
* Subject has been diagnosed with other forms of liver disease, including those with HIV and HBV co-infection, as determined by history, serological parameters, and histology when available.
* Subject has been diagnosed with a major psychiatric illness, chronic renal and/or respiratory insufficiency, intercurrent infections, treatment with sedatives within 7 days of enrollment.
* Subject shows presence of intestinal obstruction or inflammatory bowel disease, antacids or cathartics within the 12h before study start; antibiotics during 7 days before start of dosing; or treated with encephalopathy-causing agents.
* Subjects with bad vision or neurological diseases since they could have difficulty completing the neuropsychological assessments.

Phase B Inclusion Criteria

* Subject successfully participated in and continues to meet all eligibility criteria required in Phase A of the study based on completion of tests, Breath Tests, and Radiological Marker.
* Subject has a Number Connection Test score >50 sec at time of enrollment.

Phase B Exclusion Criteria

* A subject will not be eligible for inclusion in Phase B if (s)he meets any of the exclusion criteria for Phase A of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Phase A: Degree of bacterial overgrowth and its correlation with the grade of hepatic encephalopathy (if present) | 3 months
Phase B: Improvement in the psychometric scores and proportion of patients who change of HE stage | 3 months

SECONDARY OUTCOMES:
Improved Intestinal transit time | 3 months
Improvement in bacterial overgrowth | 3 months
Improved insomnia | 3 months
Improved flatulence | 3 months
Improved quality of life. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sam Sigal, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital: Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Background] Ferenci P, Lockwood A, Mullen K, Tarter R, Weissenborn K, Blei AT. Hepatic encephalopathy--definition, nomenclature, diagnosis, and quantification: final report of the working party at the 11th World Congresses of Gastroenterology, Vienna, 1998. Hepatology. 2002 Mar;35(3):716-21. doi: 10.1053/jhep.2002.31250. PMID 11870389
- [Background] Arguedas MR, DeLawrence TG, McGuire BM. Influence of hepatic encephalopathy on health-related quality of life in patients with cirrhosis. Dig Dis Sci. 2003 Aug;48(8):1622-6. doi: 10.1023/a:1024784327783. PMID 12924658
- [Background] Groeneweg M, Moerland W, Quero JC, Hop WC, Krabbe PF, Schalm SW. Screening of subclinical hepatic encephalopathy. J Hepatol. 2000 May;32(5):748-53. doi: 10.1016/s0168-8278(00)80243-3. PMID 10845661
- [Background] Groeneweg M, Quero JC, De Bruijn I, Hartmann IJ, Essink-bot ML, Hop WC, Schalm SW. Subclinical hepatic encephalopathy impairs daily functioning. Hepatology. 1998 Jul;28(1):45-9. doi: 10.1002/hep.510280108. PMID 9657095
- [Background] Amodio P, Del Piccolo F, Marchetti P, Angeli P, Iemmolo R, Caregaro L, Merkel C, Gerunda G, Gatta A. Clinical features and survivial of cirrhotic patients with subclinical cognitive alterations detected by the number connection test and computerized psychometric tests. Hepatology. 1999 Jun;29(6):1662-7. doi: 10.1002/hep.510290619. PMID 10347105
- [Background] Bustamante J, Rimola A, Ventura PJ, Navasa M, Cirera I, Reggiardo V, Rodes J. Prognostic significance of hepatic encephalopathy in patients with cirrhosis. J Hepatol. 1999 May;30(5):890-5. doi: 10.1016/s0168-8278(99)80144-5. PMID 10365817